CLINICAL TRIAL: NCT05850819
Title: Effectiveness of Gelatamp in Wound Healing After Extraction of Teeth: A Randomized Clinical Trial
Brief Title: Effectiveness of Gelatamp in Wound Healing After Teeth Extraction: A Randomized Clinical Trial
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Melaka Manipal Medical College (Other)
Responsible Party: Principal Investigator, Abdul Kalam Azad, Assistant Professor, Melaka Manipal Medical College
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MUCM/FOD/AR/B10/E C-2022(03)
Record Dates: First submitted 2023-04-29; First posted 2023-05-09 (Actual); Last update posted 2023-05-11 (Actual); Status verified 2023-05

CONDITIONS: Wound Heal

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group A (Experimental): Application of Gelatamp in the extraction socket
  Interventions: Drug: Colloidal silver gelatin sponge
- Group B (Active Comparator): Extraction socket allowed to heal without application of Gelatamp
  Interventions: Drug: Sterile gauze pack

INTERVENTIONS:
Drug: Colloidal silver gelatin sponge — Augment the extraction socket with Gelatamp
  Other Names: Gelatamp
  Arms: Group A
Drug: Sterile gauze pack — Extraction socket allowed to heal without augmentation with any material
  Arms: Group B

SUMMARY:
This study compares the effectiveness of Gelatamp for intraoral wound closure after extraction of mandibular teeth.

DETAILED DESCRIPTION:
In the interventional group, after extraction of mandibular teeth, the extraction socket will be augmented with Gelatamp. Then a gauze pack will be placed over it.

In the control group, after extraction of mandibular teeth, a gauze pack will be placed over the socket.

ELIGIBILITY:
Inclusion Criteria:

* Patients requiring extraction of mandibular teeth
* Healthy patients (ASA I) or patients with mild systemic disease but no functional limitations (ASA II)
* Patients not allergic to the drugs or anesthetics used in the study.

Exclusion Criteria:

* Patients taking medications that influences wound healing
* smokers
* Uncooperative patients
* Patients requiring extraction of grade II or III mobile teeth
* Patients requiring surgical extraction of teeth.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2023-03-30 (Actual); Study Completion 2023-03-30 (Actual)

PRIMARY OUTCOMES:
Postoperative wound healing | 7th postoperative day
  A 5 point early wound healing scale assessing wound healing after 7 postoperative days
Postoperative pain | 1st postoperative day
  A 100 mm visual analogue scale assessing postoperative pain. Possible pain scores ranges from 0 (worst pain) to 100 (worst possible pain).
Postoperative pain | 2nd postoperative day
  A 100 mm visual analogue scale assessing postoperative pain. Possible pain scores ranges from 0 (worst pain) to 100 (worst possible pain).
postoperative pain | 3rd postoperative day
  A 100 mm visual analogue scale assessing postoperative pain. Possible pain scores ranges from 0 (worst pain) to 100 (worst possible pain).
postoperative pain | 4th postoperative day
  A 100 mm visual analogue scale assessing postoperative pain. Possible pain scores ranges from 0 (worst pain) to 100 (worst possible pain).
postoperative pain | 5th postoperative day
  A 100 mm visual analogue scale assessing postoperative pain. Possible pain scores ranges from 0 (worst pain) to 100 (worst possible pain).

SECONDARY OUTCOMES:
Presence of dry socket | 3rd postoperative day
  presence of pain, foul odour, exposed bone in the extraction socket

CONTACTS AND LOCATIONS:
Overall Officials: Abdul K Azad, Principal Investigator — Melaka Manipal Medical College
Locations (1):
- Melaka Manipal Medical College, Malacca, Malaysia